CLINICAL TRIAL: NCT03498820
Title: Analgesia-Nociception Index Guided Intraoperative Remifentanil Administration Versus Standard Practice : Evaluation of Perioperative Opioid Use
Brief Title: Analgesia-Nociception Index Guided Intraoperative Remifentanil Administration Versus Standard Practice:Evaluation of Perioperative Opioid Use
Acronym: MONIDOL-ANI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P171003J
Record Dates: First submitted 2018-02-26; First posted 2018-04-17 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Pain; Anesthesia
Keywords: Analgesia-Nociception Index (ANI); General anesthesia; Opioids; Remifentanil; Pain; Monitoring
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesia Nociception Index (Experimental): Intraoperative remifentanil administration guided by the Analgesia Nociception Index
  Interventions: Device: Analgesia Nociception Index
- Usual practice (Active Comparator): Intraoperative remifentanil administration managed in standard practice
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Device: Analgesia Nociception Index — : Non invasive monitor based on heart rate variability analysis, assessing the parasympathetic nervous activity
  Other Names: ANI
  Arms: Analgesia Nociception Index
Drug: Remifentanil — intravenous short-acting opioid routinely administered during general anesthesia
  Arms: Usual practice

SUMMARY:
This study compares two groups of patients undergoing a gynecological surgey under general anesthesia: one group in which intraoperative analgesia is guided by the Analgesia-nociception index, and another group in which intraoperative analgesia is managed as in standard practice. The objective is to assess if the Analgesia Nociception Index may result in a decrease in total analgesic drugs consumption, a decrease in post-operative pain and in chronic pain development.

ELIGIBILITY:
Inclusion Criteria:

* Elective gynecological surgery under general anesthesia
* Duration of surgery 1-7 hours
* Duration of hospital stay > 24 hours

Exclusion Criteria:

* chronic pain
* chronic analgesic medication
* neurologic disease
* psychiatric disease
* history of addiction
* kidney or liver failure
* allergy to any anesthetic or analgesic drug
* BMI > 35

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | up to 7 hours after the beginning of general anesthesia
  total dose of remifentanil administered to the patient during general anesthesia

SECONDARY OUTCOMES:
Postoperative morphine consumption | obtained 24 hours after the end of general anesthesia
  total dose of morphine administered to the patient to manage postoperative pain during the first 24 hours following surgery
Persistent pain | : obtained one month after surgery
  phone interview asking the patient if she still feels pain related to the surgery
Persistent pain | Obtained three months after surgery
  phone interview asking the patient if she still feels pain related to the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nada SABOURDIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'Anesthésie-réanimation chirurgicale - Hôpital Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No